# "Predictive Value of Preoperative Evaluation in Cases of Recurrent Endometriosis" Research Informed Consent

(TİTCK-KAD-13 01.12.2019 /Ver 0.0) NCT number:2023/05/11/030

## PRIMARY RESEARCHER

Name – Evrim Ebru Kovalak
Department - Department of Obstetrics and Gynecology,
Address - University of Health Sciences, Bagcilar Training and Research
Hospital, Istanbul, Turkey
Phone - +902124404040
Email – evrimebru@yahoo.com

## PURPOSE OF STUDY

To investigate the effect of preoperative evaluation parameters in predicting recurrent disease in women who have undergone cystectomy or unilateral salpingo-oophorectomy due to endometriosis.

## **PROCEDURES**

Preoperative parameters such as biochemical parameters, cyst size and the revised American Society for Reproductive Medicine (rASRM) Scoring system will be examined for their predictive value in recurrent cases by scanning file information and computer records.

## **RISKS**

There is no risk.

## **BENEFITS**

To predict the recurrence of the disease after endometriosis surgery.

## CONFIDENTIALITY

Please do not write any identifying information.

Every effort will be made by the researcher to preserve your confidentiality including the following:

- Assigning code names/numbers for participants that will be used on all research notes and documents.
- Keeping notes, interview transcriptions, and any other identifying participant information in a locked file cabinet in the personal possession of the researcher.

| Participant's lı | nitials: |
|------------------|----------|
|------------------|----------|



Participant data will be kept confidential except in cases where the researcher is legally obligated to report specific incidents. These incidents include, but may not be limited to, incidents of abuse and suicide risk.

## **CONTACT INFORMATION**

If you have questions at any time about this study, or you experience adverse effects as the result of participating in this study, you may contact the researcher whose contact information is provided on the first page. If you have questions regarding your rights as a research participant, or if problems arise which you do not feel you can discuss with the Primary Researcher directly by telephone at 0532 4628989 or at the following email address <a href="mailto:evrimebru@yahoo.com">evrimebru@yahoo.com</a>.

## **VOLUNTARY PARTICIPATION**

Your participation in this study is voluntary. It is up to you to decide whether or not to take part in this study. If you decide to take part in this study, you will be asked to sign a consent form. After you sign the consent form, you are still free to withdraw at any time and without giving a reason. Withdrawing from this study will not affect the relationship you have, if any, with the researcher. If you withdraw from the study before data collection is completed, your data will be returned to you or destroyed.

Note: Please delineate the "Consent" section of the Informed Consent Form by drawing a line across the page (like this - Example). This delineation is important because the consent form grammar shifts from second person to first person, as shown in the example.

## CONSENT

I have read and I understand the provided information and have had the opportunity to ask questions. I understand that my participation is voluntary and that I am free to withdraw at any time, without giving a reason and without cost. I understand that I will be given a copy of this consent form. I voluntarily agree to take part in this study.

| Participant's Signature | Date |
|-------------------------|------|
| Researcher's Signature | Date |
| - | |

| P | artici | pant's | Initials: |
|---|--------|--------|-----------|

